CLINICAL TRIAL: NCT02331199
Title: Comparison Between Amniotic Fluid Lamellar Body Count and Fetal Pulmonary Artery Doppler Indices in Predicting Fetal Lung Maturity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: preterm 1
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Preterm Labour
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- preterm labour (Experimental): 200 women with preterm prelabour ruptured membranes or undergoing preterm CS
  Interventions: Device: Amniotic fluid lamellar body count; Device: Fetal pulmonary artery Doppler

INTERVENTIONS:
Device: Amniotic fluid lamellar body count — The LBC (the unit of measurement is number of lamellar bodies counted per microliter of amniotic fluid) will be determined using the platelet channels on the Hematology Flow Cytometer.
  Other Names: Amniotic fluid lamellar body count will be measured
Device: Fetal pulmonary artery Doppler — A fetal pulmonary artery Doppler will be performed using color Doppler ultrasound. Doppler flow velocity measurements, including systolic/diastolic ratio, pulsatility index, resistance index, and acceleration-time/ejection-time ratio using spectral Doppler ultrasound.

SUMMARY:
The investigators will study 200 women with singleton pregnancies presented with prelabor preterm rupture of membranes or undergoing cesarean section (CS). Amniotic fluid lamellar body count (LBC) and fetal pulmonary artery Doppler will be done to all women. LBC and fetal pulmonary artery Doppler will be correlated with fetal outcome

DETAILED DESCRIPTION:
Neonatal respiratory distress syndrome (RDS) remains a major cause of neonatal morbidity and mortality. A recent epidemiologic study in the United States estimates that there are 80,000 cases of neonatal RDS each year, resulting in 8500 deaths and hospital costs in excess of $4.4 billion.

A number of biochemical tests have been developed to predict the risk of RDS and assist obstetric care providers in delivery timing. Amniotic fluid lamellar body count (LBC) is an important biophysical test, based on measuring the concentration of pulmonary surfactant in amniotic fluid. It can be effectively used to assess fetal lung maturity. A noninvasive test for fetal lung maturity (FLM) would be useful to minimize the need for invasive testing and would be more acceptable to women. Fetal pulmonary artery Doppler waveform acceleration/ejection time may provide a noninvasive means of determining fetal lung maturity with relatively acceptable levels of sensitivity, specificity, and predictive values.

The investigators will study 200 women with singleton pregnancies presented with prelabor preterm rupture of membranes or undergoing cesarean section (CS). Amniotic fluid lamellar body count (LBC) and fetal pulmonary artery Doppler will be done to all women. LBC and fetal pulmonary artery Doppler will be correlated with fetal outcome.

Quantitative data will be statistically represented in terms of mean ± standard deviation (± SD) while categorical data will be represented as frequency and percentage. Comparison of quantitative data will be done using Mann Whitney U test for independent samples while categorical data will compared using Chi squared test or Fisher exact test when appropriate. A probability value (p value) less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies without any major congenital anomalies.
* Gestation between 32-36 weeks
* Women presenting preterm pre-labour ruptured membranes or undergoing a cesarean section.

Exclusion Criteria:

* Patients with major fetal anomalies.
* Bloody or meconium stained amniotic fluid
* preexisting maternal medical conditions (eg, diabetes, renal disease, hypertensive disorders, vaginal bleeding

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory distress syndrome (RDS) | 1 day after delivery
  RDS will be diagnosed clinically by the presence of tachypnea, working respiratory muscles, expiratory grunt, and chest x-ray.

SECONDARY OUTCOMES:
Need for incubation | 1 day after delivery
  It will be recorded if the pediatrician decides to incubate the neonate. The reason for incubation e.g. ventilation, hypoxia, ischemia will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al Galaa maternity fospital, Cairo
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] AVERY ME, MEAD J. Surface properties in relation to atelectasis and hyaline membrane disease. AMA J Dis Child. 1959 May;97(5, Part 1):517-23. doi: 10.1001/archpedi.1959.02070010519001. No abstract available. PMID 13649082
- [Background] Dubin SB. Characterization of amniotic fluid lamellar bodies by resistive-pulse counting: relationship to measures of fetal lung maturity. Clin Chem. 1989 Apr;35(4):612-6. PMID 2702746
- [Background] Neerhof MG, Dohnal JC, Ashwood ER, Lee IS, Anceschi MM. Lamellar body counts: a consensus on protocol. Obstet Gynecol. 2001 Feb;97(2):318-20. doi: 10.1016/s0029-7844(00)01134-0. PMID 11165603